CLINICAL TRIAL: NCT03356470
Title: Pilot Study of Biomarkers of Response to Immune Checkpoint Blockade in Metastatic Melanoma
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2017-0046; 2017-0046 (Other: Institutional Review Board); P30CA014520 (NIH); A534260 (Other: UW Madison); SMPH\MEDICINE\HEM-ONC (Other: UW Madison); Protocol Version 6/19/2019 (Other: UW Madison)
Record Dates: First submitted 2017-11-22; First posted 2017-11-29 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2022-07

CONDITIONS: Melanoma
Keywords: melanoma; antimelanoma T cells
MeSH Terms: conditions — Melanoma | interventions — alovudine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- FLT/PET + biopsy: F-FDG and FLT PET/CT imaging will be obtained prior to anti-cancer treatment and 10-12 weeks after starting treatment with anti-PD-1 antibody.
  Interventions: Other: F-FDG PET/CT

INTERVENTIONS:
Other: F-FDG PET/CT — F-FLT PET uses a thymidine analogue that accumulates in proliferating tissue. Proliferating tissue could include malignant lesions or immune cells. In this study, FLT PET/CT will be utilized as a molecular imaging tool to detect immune activation after administration of immune checkpoint blockade with pembrolizumab or nivolumab.
  Other Names: 3'-Deoxy-3'-[18F]Fluorothymidine (FLT) PET/CT

SUMMARY:
This study uses molecular imaging and novel immune monitoring to identify a biomarker of response for melanoma patients receiving immunotherapy with anti-PD-1 immunotherapy. Prior to treatment, FDG and FLT PET/CT will be obtained, together with blood and tumor biopsies from each patient. A follow-up FDG and FLT PET/CT will be obtained, together with blood and tumor biopsies, 10-12 weeks after starting treatment with anti-PD-1 antibody. Additional tumor biopsies and blood samples for immune monitoring will be obtained 4-6 weeks after starting treatment with anti-PD-1 antibody as well as 16-18 weeks after starting anti-PD-1 treatment for patients still receiving anti-PD-1 antibody at that time.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a metastatic melanoma diagnosis (stage IV) for which treatment with nivolumab or pembrolizumab, either alone or in combination with other therapies, is planned. No additional laboratory testing is needed for the imaging in this study apart from the standard laboratory testing routinely obtained for treatment with nivolumab or pembrolizumab, either alone or in combination with other therapies.
* Participants must have at least 2 subcutaneous or lymph node melanoma metastases that are 2 cm in greatest diameter and are amenable to being biopsied in clinic without requiring image-guidance.
* Participants must be able to provide informed consent
* Women of childbearing potential must be willing to use effective contraception as discussed with their oncologist while participating in this study.

Exclusion Criteria:

* Not able to receive treatment with either nivolumab or pembrolizumab.
* Women of child-bearing potential must have a negative serum or urine pregnancy test within 7 days of the first study FLT PET/CT and must not be breast feeding for the duration of study participation.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Up to 4 metastatic melanoma patients will be recruited from the University of Wisconsin (UW) Carbone Cancer Center (CCC) Melanoma Clinic located in the UW-Hospital and Clinics.
Sampling Method: Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2017-11-02 (Actual); Primary Completion 2022-06-17 (Actual); Study Completion 2022-06-17 (Actual)

PRIMARY OUTCOMES:
Correlation of baseline of response and antitumor response | Anticipated at one-year after last patient enrolled, around Sept 2019
  To correlate baseline and post-treatment molecular imaging biomarkers of response to immunotherapy with anti-PD-1 with antitumor response based on analysis of the FDG-to-FLT PET/CT ratio in melanoma patients

SECONDARY OUTCOMES:
Correlation of in vivo clonally amplified T cells to FDG PET uptake in melanoma tumors | Anticipated at one-year after last patient enrolled, around Sept 2019
  To correlate in vivo clonally amplified T cells in blood that traffic to tumor to FDG PET uptake in melanoma tumors following treatment with anti-PD-1
To correlate histologic and molecular markers of antitumor response to FLT PET uptake in melanoma tumors following treatment with anti-PD-1 | Anticipated at one-year after last patient enrolled, around Sept 2019
  To correlate histologic and molecular markers of antitumor response to FLT PET uptake in melanoma tumors following treatment with anti-PD-1

CONTACTS AND LOCATIONS:
Overall Officials: Mark Albertini, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Carbone Cancer Center, Madison, Wisconsin, United States

REFERENCES:
- See also: University of Wisconsin Carbone Cancer Center Home — https://cancer.wisc.edu